CLINICAL TRIAL: NCT02362841
Title: Assessment of the Evolutions of Transcutaneous CO2 With the Modification of Blood Flow During On-pump Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Pirracchio Romain, Dr, European Georges Pompidou Hospital
Other Study IDs: HEGP-SAR-001
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: PtCO2, Extracorporeal Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There are no available criteria for determining the optimal flow rate and mean arterial pressure level in patients under cardiopulmonary bypass (CPB). Transcutaneous carbon dioxide tension (PtCO2) has been proposed for microcirculation monitoring and it could be useful for guiding hemodynamic optimization under CPB. The goal of this exploratory study was to determine the factors that influence PtCO2 variations during CPB.

DESIGN: Cutaneous ear lobe CO2 tension was monitored along with hemodynamic parameters every 10 minutes during CPB, until aortic unclamping. SETTING: French university teaching hospital PARTICIPANTS: Patients scheduled for cardiac surgery requiring CPB were prospectively included.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cardiac surgery under cardiac arrest and cardiopulmonary bypass were prospectively included in the present observational study conducted at a French teaching hospital.

Exclusion Criteria:

* The exclusion criteria were: age <18, pregnancy, septic or emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery under cardiac arrest and cardiopulmonary bypass were prospectively included in the present observational study conducted at a French teaching hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PtCO2 | intraoperative value